CLINICAL TRIAL: NCT00080431
Title: An Open Label Trial to Assess Safety and Tolerability of Daclizumab in HIV-Infected Individuals
Brief Title: Daclizumab to Treat HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040149; 04-I-0149
Record Dates: First submitted 2004-03-30; First posted 2004-03-31 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-12-28

CONDITIONS: HIV Infections
Keywords: Reservoir; Viral Load; Immunosuppression; Activation; Latency; HIV; HAART; Immunosuppressive Drug; Viral Reservoirs
MeSH Terms: conditions — HIV Infections | interventions — Daclizumab

INTERVENTIONS:
Drug: Daclizumab

SUMMARY:
This study will examine the safety and effectiveness of daclizumab (also called Zenapax or anti-CD25) in reducing viral replication in patients with HIV infection. Although HAART, an intensive anti-HIV treatment regimen, can suppress HIV in blood below the limit of detection, it cannot completely eradicate the virus. This study will focus on the effectiveness of daclizumab in further reducing viral replication in patients with low viral counts. The Food and Drug Administration approved daclizumab in 1997 for preventing kidney transplant rejection, and it has also been studied in people with an eye infection called uveitis. The drug works by binding to a protein on T cells (white blood cells of the immune system) called CD25. This prevents another protein, called interleukin-2 (IL-2), from binding to this site, thus preventing a series of events that normally results in inflammation.

Patients between 18 and 65 years of age with HIV infection who have stable HIV levels at less than 30,000 copies/mL of blood and CD4 T cell counts higher than 400 cells/cmm may be eligible for this study. Patients who have taken drugs that affect the immune system, such as IL-2 and interferon, in the past 5 years may not participate. Candidates are screened with a comprehensive medical examination, including physical examination and laboratory studies. X-rays, consultations, and biopsies are done only if medically indicated.

Participants will undergo the following tests and procedures:

* Daclizumab therapy: Patients receive daclizumab as a 25-minute infusion through an intravenous catheter (plastic tube placed in a vein) at the NIH Clinical Center outpatient clinic. A total of three doses of drug are given. The first dose is given on study day 1, the second dose is given 2 weeks later, and the third dose is given 4 weeks later. Patients are observed for at least 1 hour after each infusion before being discharged from the clinic.
* Follow-up visits: Patients return to the outpatient clinic every 2 weeks while they are on medication and then every month until 3 months after the final dose to evaluate their infection status, response to therapy, and medication side effects. The visits include a physical examination, blood draws, and possibly x-rays, if medically indicated.
* Apheresis: Patients undergo apheresis, a procedure for collecting large amounts of white blood cells, three times during the study - once before starting daclizumab therapy, 4 weeks after beginning therapy, and 12 weeks after beginning therapy. For apheresis, blood is removed through a needle in the vein of one arm and spun in a machine that separates it into its components. The white blood cells and plasma are removed, and the red cells and platelets are re-infused either through the same needle or through a needle in a vein in the other arm.

DETAILED DESCRIPTION:
The purpose of this protocol is to evaluate the safety and tolerability of an immunosuppressive agent, daclizumab, in HIV-infected adults. HIV-infected individuals with levels of plasma viremia below 30,000 copies/mL will receive daclizumab for one month. Various immunologic and virologic laboratory studies addressing the state of cellular activation and toxicity data will be collected post-enrollment. The primary study risks include factors associated with immunosuppression and fluctuation on HIV viral levels. Subjects will be compensated for participation in this study. Total enrollment for the study will be a maximum of 10 subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Documentation of HIV-1 infection by licensed ELISA test and confirmed by a Western Blot.
  2. Demonstration of control of HIV viremia below the 30,000 copies/mL with a variability of less than 0.5 log of baseline two times within a week and a stable viral load for the previous 3 months. Patient may or may not be on HAART.
  3. Patients with CD4 cell count greater than 400 cells/mm(3) at time of screening visit. A variability of 10% between two values is acceptable for values below 400.
  4. Ability to sign informed consent and willingness to comply with the study requirements and clinic policies.
  5. Age 18-65 years.
  6. Willingness to travel to the NIH every 2-4 weeks
  7. Need to have a primary doctor who will be taking care of the patients for their HIV infection.
  8. Willingness of both women and men to use an effective means of birth control while receiving treatment through this study and 3 months following treatment. Appropriate birth control includes barrier methods, sterilization, and birth control pills.
  9. Willing to designate a person for durable power of attorney on the NIH form for medical research and medical care purposes at the NIH Clinical Center.
  10. Willing to undergo genetic testing for HLA and willing to have samples stored for future research

EXCLUSION CRITERIA:

1. Patients who are pregnant or who are nursing infants will not be eligible. Women of child-bearing potential must have a negative pregnancy test on the day of study entry.
2. Acute or chronic liver disease, history of alcohol abuse or drug abuse that would interfere with participation in the clinical trial.
3. History of any malignant neoplasm except in situ anogenital carcinoma, adequately treated basal or squamous cell carcinoma of the skin, or solid tumors treated with curative therapy and disease free for at least 5 years.
4. History of bladder cancer.
5. Previous treatment with daclizumab.
6. Inability to comply with study guidelines.
7. Hemocytopenia: platelet count less than 80,000/mm(3), absolute neutrophil count less than 1500/mm(3), hematocrit less than 30% (in the absence of gastrointestinal bleeding or hemolytic anemia).
8. ALT/AST greater than 5 times the upper limit of normal, PT INR greater than 2 times the upper limit of normal, creatinine greater than 1.5 times the upper limit of normal.
9. Concurrent use of any other immunosuppressive therapy including systemic steroids for a duration of six weeks or more six months prior to enrollment.
10. History of use of the immunomodulatory agent such as IL-2 or interferon within the last 5 years.
11. Known allergy to murine proteins.
12. Medical illness that in the opinion of the investigator might confound results or interfere with the subject's ability to participate in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2004-03-26; Study Completion 2007-12-28

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wong JK, Hezareh M, Gunthard HF, Havlir DV, Ignacio CC, Spina CA, Richman DD. Recovery of replication-competent HIV despite prolonged suppression of plasma viremia. Science. 1997 Nov 14;278(5341):1291-5. doi: 10.1126/science.278.5341.1291. PMID 9360926